CLINICAL TRIAL: NCT00434161
Title: A Double-Blind, Randomized, Placebo-controlled Study of Two Different Schedules of Palifermin for Reduction in Severity of Oral Mucositis in Subjects With Multiple Myeloma Receiving Melphalan Followed by Autologous Blood Stem Cell Transplantation
Brief Title: A Study of Palifermin for the Reduction of Oral Mucositis in Subjects With Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 20050219; NCT00964925 (obsolete NCT alias)
Record Dates: First submitted 2007-02-08; First posted 2007-02-12 (Estimated); Results first posted 2015-03-10 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Multiple Myeloma
Keywords: Palifermin; KGF; Clinical Trial; Oncology; Oral Mucositis; Multiple Myeloma; Cataract
MeSH Terms: conditions — Multiple Myeloma; Neoplasms; Stomatitis; Cataract | interventions — Fibroblast Growth Factor 7

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Palifermin before only (Active Comparator): Subjects received palifermin before-high dose chemotherapy (total 3 doses) and matched placebo after-high dose chemotherapy (total 3 doses)
  Interventions: Drug: Palifermin before only
- Placebo (suger pill) (Placebo Comparator): Subjects received matched placebo before- and after-high dose chemotherapy
  Interventions: Drug: Placebo
- Palifermin before and after (Active Comparator): Subjects received palifermin before- and after-high dose chemotherapy (total of 6 doses)
  Interventions: Drug: Palifermin before and after

INTERVENTIONS:
Drug: Palifermin before only — One bolus IV injection at 60 μg/kg/day, on Days 6, 5 & 4 days before-high dose chemotherapy and one bolus IV injection at 60 μg/kg/day of matched placebo on days 0, 1 & 2 days after-high dose chemotherapy. Minimum of 4 days between before-chemotherapy and after-transplantation dosing.
  Other Names: Kepivance
  Arms: Palifermin before only
Drug: Placebo — One bolus IV injection at 60 μg/kg/day of matched placebo on Days 6, 5 & 4 (before-high dose chemotherapy) and on Days 0, 1 & 2 (after-high dose chemotherapy).
  Minimum of 4 days between pre-chemotherapy and post-transplantation dosing.
  Arms: Placebo (suger pill)
Drug: Palifermin before and after — One bolus IV injection at 60 μg/kg/day, on Days 6, 5 & 4 (before-high dose chemotherapy) and on Days 0, 1 & 2 (after-high dose chemotherapy).
  Minimum of 4 days between before-chemotherapy and after-transplantation dosing.
  Other Names: Kepivance
  Arms: Palifermin before and after

SUMMARY:
The purpose of this study was to evaluate the efficacy and effect of palifermin on the incidence of oral mucositis in subjects with multiple myeloma receiving Melphalan followed by autologous peripheral blood stem cell transplantation. Amendment 01 (April 07) introduced three cataract assessments to be carried out at Screening, Month 6 and Month 12 in response to FDA and EMEA follow up measures.

DETAILED DESCRIPTION:
This was a double-blind, placebo-controlled, randomized, multicenter Phase IIIb study of palifermin given before and after dose chemotherapy (total 6 doses) or before dose chemotherapy only (total 3 doses), in subjects with Multiple Myeloma (MM)receiving high dose melphalan (chemotherapy), in a 1-day schedule, followed by autologous Peripheral Blood Stem Cell Transplantation (PBSCT).

All subjects were to be followed for disease progression, second primary tumors, additional malignancies and survival for up to 10 years.

Planned: 275 subjects, in fact, 281 subjects were randomized. Randomized: 115 subjects to palifermin pre/post-CT, 109 subjects to palifermin pre-CT and 57 subjects to placebo Analyzed: 281 subjects in the full analysis set, 277 subjects in the safety subset.

Efficacy Oral cavity assessment, patient reported outcome (PRO) questionnaires (Oral Mucositis Daily Questionnaire [OMDQ], Functional Assessment of Cancer Therapy Esophageal [FACT-E], European Quality of Life Utility Scale [EQ 5D], Mucositis Chronic Symptoms Questionnaire [MCSQ]).

Safety Physical examination (including body temperature), concomitant medications, transfusions, vital signs, laboratory assessments (hematology, chemistry), cataract assessments, adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

* Multiple myeloma (MM) subjects scheduled to receive high-dose Melphalan in a one day schedule followed by autologous peripheral blood progenitor cell (PBSCT)
* Body Mass Index (BMI) ≤ 35
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2, or an ECOG status of 3 if the reason for a status of 3 is exclusively due to MM (e.g. pathological fracture)
* Functional hematopoietic, hepato-renal and pulmonary systems
* Subjects at minimum with a baseline best corrected visual acuity (BCVA) of 20/40, (6/12 or 0.5 on the decimal scale) or better using the ETDRS chart in one eye
* Subject at minimum with one eye with a natural, intact lens
* Subject who has a LOCS III score at baseline of P < 1.0, C < 2.0 and NO < 2.0 in at least one eye
* Women in child bearing potential must have a negative pregnancy test

Exclusion Criteria:

* Presence or history of any other malignancy (other than curatively treated basal cell or squamous cell carcinoma of the skin, in situ cervical carcinoma, or other surgically cured malignancy, without evidence of disease for > 3 years
* Prior autologous or allogeneic transplants
* Prior treatment with palifermin, or other fibroblast or keratinocyte growth factors
* Receiving dialysis
* History of cataract surgery in both eyes
* Incapable of being responsive to mydriatic agents
* History of other ocular disease (e.g., macular degeneration, glaucoma, corneal disease) that would make assessment of visual status difficult
* Subject is scheduled to undergo cataract surgery
* Subject with any disease, that in the opinion of the ophthalmologist, could adversely effect the subject's vision during the course of the study
* Currently active oral mucositis infection
* Positive for HIV, hepatitis B or C
* Subject is unable or unwilling to follow with study procedures
* Subject is pregnant or is breast feeding
* Subject has not agreed to use adequate contraceptive precautions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2006-12; Primary Completion 2009-03 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Timdahl, MD, Study Director — Swedish Orphan Biovitrum AB; Dietger Niederwieser, Professor, Principal Investigator — Universitatsklinikum Leipzig, Leipzig, Germany
Locations (1):
- Universitatsklinikum Leipzig, Leipzig, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Palifermin Before Only: Subjects to receive palifermin before-high dose chemotherapy (total 3 doses) and matched placebo after-high dose chemotherapy (total 3 doses). Daily dose of intravenous (IV) 60 µg/kg/day of palifermin as 1 bolus IV injection on Days -6, 5 and -4 before high dose chemotherapy and placebo on Days 0, 1 and 2 after high dose chemotherapy.
- Placebo: Subjects to receive matched placebo before- and after-high dose chemotherapy (total of 6 doses). Daily dose of intravenous (IV) 60 µg/kg/day of placebo as 1 bolus IV injection on Days -6, 5 and -4 before high dose chemotherapy and on Days 0, 1 and 2 after high dose chemotherapy.
- Palifermin Before and After: Subjects to receive palifermin before- and after-high dose chemotherapy (total of 6 doses). Daily dose of intravenous (IV) 60 µg/kg/day of palifermin as 1 bolus IV injection on Days -6, 5 and -4 before high dose chemotherapy and on Days 0, 1 and 2 after high dose chemotherapy
Period: Overall Study
Arm/Group | Palifermin Before Only | Placebo | Palifermin Before and After
Started | 109 | 57 | 115
Completed | 99 | 54 | 104
Not Completed | 10 | 3 | 11
Not completed — Adverse Event | 5 | 1 | 4
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Death | 1 | 0 | 1
Not completed — Non-Compliance | 1 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 3
Not completed — Logistical error study assessments | 1 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Palifermin Before Only: Subjects to receive palifermin before-high dose chemotherapy (total 3 doses) and matched placebo after-high dose chemotherapy (total 3 doses)
- Placebo: Subjects to receive matched placebo before- and after-high dose chemotherapy
- Palifermin Before and After: Subjects to receive palifermin before- and after-high dose chemotherapy (total of 6 doses)
- Total: Total of all reporting groups
Arm/Group | Palifermin Before Only | Placebo | Palifermin Before and After | Total
Number analyzed (Participants) | 109 | 57 | 115 | 281
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 90 | 49 | 100 | 239
  >=65 years | 19 | 8 | 15 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (8.4) | 57.1 (7.0) | 56.1 (7.5) | 56 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 24 | 52 | 126
  Male | 59 | 33 | 63 | 155
Region of Enrollment [Number; unit: participants]
  Germany | 16 | 9 | 23 | 48
  Hungary | 22 | 9 | 16 | 47
  France | 15 | 10 | 16 | 41
  Austria | 16 | 5 | 9 | 30
  Belgium | 8 | 1 | 11 | 20
  Czech Republic | 7 | 4 | 7 | 18
  Italy | 4 | 4 | 9 | 17
  Switzerland | 4 | 5 | 6 | 15
  United Kingdom | 4 | 2 | 5 | 11
  Finland | 3 | 3 | 4 | 10
  Netherlands | 4 | 1 | 5 | 10
  Ireland | 2 | 2 | 3 | 7
  Sweden | 2 | 1 | 1 | 4
  Denmark | 2 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Maximum Severity of Oral Mucositis (World Health Organization (WHO) Grades 0/1, 2, 3, or 4)
Description: For the primary efficacy endpoint maximum severity of Oral Mucositis (OM) was assessed, the number of participants who had the different severity. To assess severity of OM, a 5-grade WHO scale (0, 1, 2, 3, or 4) was used.
  0 = no findings or erythema only, 1= soreness present with or without erythema, 2=ulcers present but able to take solid food, 3 =ulcers present and only able to take liquids, 4 =ulcers present/not able to take anything orally.
Time Frame: at Day 32
Population: Full analysis set that includes all randomized subjects, and was used to compare treatment effects for all efficacy endpoints. This set of subjects was analyzed according to their randomized treatment assignment.
Measure: Number; unit: Participants
Groups:
- Palifermin Before Only: Subjects to receive palifermin before-high dose chemotherapy and matched placebo after-high dose chemotherapy
- Palifermin Before and After: Subjects to receive palifermin before- and after-high dose chemotherapy
Arm/Group | Palifermin Before Only | Placebo | Palifermin Before and After
Number analyzed (Participants) | 109 | 57 | 115
Participants
  WHO grade 0/1 or 2 | 79 | 36 | 68
  WHO grade 3 or 4 | 26 | 21 | 44
  Unknown | 4 | 0 | 3
Statistical Analysis 1: Comparison: Placebo vs Palifermin Before and After; The null hypothesis was that the severity distribution for OM was identical for the placebo and each of the two palifermin groups, and the alternative hypothesis was that palifermin resulted in a shift in the distribution to less severe mucositis than placebo. A total of 275 subjects would give at least 95% power, with a 2.5% type I error rate for each comparison to detect an odds ratio of at least 3.5 between the placebo group and each of the two palifermin groups; Test type: Superiority or Other; p = 0.188, Proportional odds model — A 2.5% type I error rate for each comparison gives an overall type I error rate of 5%; The proportional odds model including the randomization factors as covariates was used for the primary endpoint, maximum severity of OM; Odds Ratio (OR) = 0.679, 97.5% CI 2-sided [0.351 to 1.313] — The odds ratio was defined to be the odds of a subject receiving placebo experiencing OM divided by the odds of a subject receiving palifermin developing OM
Statistical Analysis 2: Comparison: Palifermin Before Only vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.468, Proportional odds model — A 2.5% type I error rate for each comparison gives an overall type I error rate of 5%; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.242, 97.5% CI 2-sided [0.635 to 2.431] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Incidence Ulcerative Mucositis (WHO Grades 2, 3, and 4)
Description: The incidence of ulcerative mucositis WHO grades 2, 3, and 4. Measured the number of participants who had WHO grades 2, 3, and 4:
  2=ulcers present but able to take solid food, 3=ulcers present and only able to take liquids, 4=ulcers present/not able to take anything orally.
Time Frame: at Day 32
Population: Full analysis set that includes all randomized subjects (total 281 subjects), and was used to compare treatment effects for all efficacy endpoints. This set of subjects was analyzed according to their randomized treatment assignment.
Measure: Number; unit: participants
Arm/Group | Palifermin Before Only | Placebo | Palifermin Before and After
Number analyzed (Participants) | 109 | 57 | 115
participants
  Incidence (n): yes | 56 | 33 | 79
  Incidence (n): No | 49 | 24 | 33
  Incidence (n): unknown | 4 | 0 | 3
Statistical Analysis 1: Comparison: Placebo vs Palifermin Before and After; Test type: Superiority or Other; p = 0.245, Cochran-Mantel-Haenszel — For secondary endpoints the type I error was protected by using the Hochberg procedure. The reported p-values are adjusted by the Hochberg procedure; Risk Difference (RD) = 13.262, 97.5% CI 2-sided [-4.303 to 30.828]
Statistical Analysis 2: Comparison: Palifermin Before Only vs Placebo; Test type: Superiority or Other; p = 0.806, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Risk Difference (RD) = -2.014, 97.5% CI 2-sided [-20.519 to 16.491]

3. Secondary Outcome: Duration of Ulcerative Mucositis (WHO Grades 2, 3, and 4)
Description: The duration of ulcerative mucositis measured the number of days the participants had different WHO grades 2, 3, and 4:
  2=ulcers present but able to take solid food, 3 =ulcers present and only able to take liquids, 4 =ulcers present/not able to take anything orally. Patients that did not have any ulcerative mucositis were given a value of 0 days.
Time Frame: at Day 32
Population: as for outcome 2
Measure: Mean (Full Range); unit: Days
Arm/Group | Palifermin Before Only | Placebo | Palifermin Before and After
Number analyzed (Participants) | 109 | 57 | 115
Days | 4.78 (6.13) [0 to 32] | 4.98 (5.95) [0 to 25] | 7.38 (6.82) [0 to 27]
Statistical Analysis 1: Comparison: Placebo vs Palifermin Before and After; A type I error rate was protected by using the Hochberg procedure to adjust for multiple testing. Palifermin was not to be declared to be statistically superior to placebo with respect to secondary efficacy endpoints unless the primary endpoint was statistically significant in favor of palifermin; Test type: Superiority or Other; p = 0.095, van Elteren test — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 2.409, 97.5% CI 2-sided [0.070 to 4.748], Standard Deviation 6.82
Statistical Analysis 2: Comparison: Palifermin Before Only vs Placebo; Test type: Superiority or Other; p = 0.806, van Elteren test — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.213, 97.5% CI 2-sided [-2.575 to 2.150], Standard Deviation 6.13

4. Secondary Outcome: The Area Under the Curve (AUC) Was Calculated From the Patient-reported Outcome Mouth and Throat Soreness (MTS) Score.
Description: The mean daily scores were calculated using the subject daily assessment of Patient-reported mouth and throat soreness (MTS) on the 5 point scale with higher values in MTS indicating a worse self assessed MTS. A 5-grade WHO scale (0, 1, 2, 3, or 4). 0=no findings or erythema only, 1=soreness present with or without erythema, 2=ulcers present but able to take solid food, 3=ulcers present and only able to take liquids, 4=ulcers present/not able to take anything orally. The incidence of ulcerative mucositis WHO grades 2, 3, and 4. Measured the number of participants who had WHO grades 2, 3, and 4:
  2=ulcers present but able to take solid food, 3=ulcers present and only able to take liquids, 4=ulcers present/not able to take anything orally. The area under the curve were calculated at the time points; Day(D)-2, up to Day 32.
Time Frame: at Day 32
Measure: Mean (Standard Deviation); unit: units on a scale * days
Arm/Group | Palifermin Before Only | Placebo | Palifermin Before and After
Number analyzed (Participants) | 109 | 57 | 115
units on a scale * days | 29.82 (45.04) | 24.55 (32.35) | 39.97 (52.90)
Statistical Analysis 1: Comparison: Placebo vs Palifermin Before and After; For the secondary endpoints, the type I error rate was protected by using the Hochberg procedure to adjust for multiple testing16. Palifermin was not to be declared to be statistically superior to placebo with respect to secondary efficacy endpoints unless the primary endpoint was statistically significant in favor of palifermin; Test type: Superiority or Other; p = 0.142, van Elteren test — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 15.436, 97.5% CI 2-sided [-1.542 to 32.415]
Statistical Analysis 2: Comparison: Palifermin Before Only vs Placebo; Test type: Superiority or Other; p = 0.806, van Elteren test — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 5.331, 97.5% CI 2-sided [-11.820 to 22.482]

5. Secondary Outcome: Incidence of Cataract Development or Progression (Change of ≥0.3 in Lens Opacities Classification System III (LOCS III Score)) at Month 6.
Description: Number of participants from the primary cataract subset showing an increase from baseline of >= 0.3 in the Lens Opacities Classification System III (LOCS III score). The LOCS III is a standard system used for grading and comparison of cataract severity and type. The ophthalmologist trained in LOCS III uses a slit lamp for examining the lens of the eye. The classification evaluates four features: posterior subcapsular cataract(P),cortical cataract(C),nuclear opalescence(NO) and nuclear color(NC). NO and NC are graded on a decimal scale of 0.1 to 6.9, based on a set of 6 standardized photographs. C and P are graded on a decimal scale of 0.1 to 5.9, based on a set of 5 standardized photographs each. In the current study, cataract development or progression was defined as an increase from baseline of ≥ 0.3 on any of the three features P, C or NO (NC is of less importance and has not been analysed further in this study).
Time Frame: 6 Months
Population: Of the 281 subjects who participated in the acute phase of the study a total of 101 subjects study were eligible for participation in the cataract assessment procedures, 22 in the placebo group and 79 in the palifermin group. Number of patients with non-missing values at Months 6; were 17 in the placebo group and 53 in the palifermin group.
Measure: Number; unit: participants
Groups:
- Palifermin: Subjects to receive Before- and After chemotherapy, and Before chemotherapy only
Arm/Group | Placebo | Palifermin
Number analyzed (Participants) | 22 | 79
participants
  Yes | 6 | 23
  No | 11 | 30
  Missing | 5 | 26
Statistical Analysis 1: Comparison: Placebo vs Palifermin; Test type: Superiority or Other; According to statistical analysis plan it was not planned to calculate any P-Value; Risk Difference (RD) = 5.88, 95% CI 2-sided [-21.669 to 33.43]

6. Secondary Outcome: Incidence of an Increase Posterior Subcapsular Cataract (P), Cortical Cataract (C) and Nuclear Opalescence (NO) at Month 6 and 12
Description: To assess the effect of palifermin on the incidence of cataract development or progression at Month 6 and Month 12 based on an increase of ≥ 0.3 in the Lens Opacities Classification System (LOCS III) score for Posterior (P), Cortical Cataract (C) and Nuclear Opalescence (NO).
  For Subcapsular cataract (P), Cortical Cataract (C) and Nuclear Opalescence (NO): at month 6 and 12 adjusted difference of rate of cataract, Palifermin - Placebo were used and the confidence interval were calculated on the adjusted difference.
Time Frame: at Month 6 and Month 12
Population: 281 subjects participated in the acute phase study of those 101 subjects were eligible for the cataract assessment study, 22 placebo and 79 palifermin. Month 6: 69 completed (17/22 [77.3%] in the placebo, 52/79 [65.8%] in the palifermin. Month 12: 66 completed (14/22 [63.6%] in the placebo, 52/79 [65.8%] in the palifermin group.
Measure: Number; unit: participants
Arm/Group | Placebo | Palifermin
Number analyzed (Participants) | 22 | 79
participants
  P month 6 - Yes | 0 | 5
  P, month 6 - No | 17 | 47
  P, month 12 - Yes | 1 | 13
  P, month 12 - No | 13 | 39
  C month 6 - Yes | 3 | 9
  C, month 6 - No | 14 | 43
  C, month 12 - Yes | 2 | 13
  C, month 12 - No | 12 | 39
  NO month 6 - Yes | 3 | 19
  NO month 6 - No | 14 | 33
  NO month 12 - Yes | 4 | 20
  NO month 12 - No | 10 | 32
  P, C and NO, month 6 - Subjects who discontinued | 5 | 27
  P, C and NO, month 12 - Subjects who discontinued | 8 | 27

7. Secondary Outcome: Change From Baseline in Posterior Subcapsular (P), Cortical (C) Cataract and Nuclear Opalescence (NO) on the Lens Opacities Classification System III (LOCS III) Scale at Months 6.
Description: To study the change in cataract from baseline visit to months 6, three cataract main types: nuclear, cortical and posterior subcapsular measured on the Lens Opacities Classification System III (LOCS III) Scale.
  To assess the effect of palifermin on the incidence of cataract development or progression at Month 6 and Month 12 based on an increase of ≥ 0.3 in theLOCS III score for Posterior Subcapsular cataract (P), Cortical Cataract (C) and Nuclear Opalescence (NO).
  The LOCS III is a standard system used for grading and comparison of cataract severity and type. The ophthalmologist uses a slit lamp for examining the lens of the eye. The classification evaluates: P,C and NO. NO is graded on a decimal scale of 0.1 to 6.9, based on a set of 6 standardized photographs. C and P are graded on a decimal scale of 0.1 to 5.9, based on a set of 5 standardized photographs each.
Time Frame: Months 6
Population: All subjects in the acute phase study were also assessed for their eligibility for cataract assessment procedures according to predefined criteria. If a subject was not eligible for cataract assessment procedures, the subject could still have been eligible for inclusion in the study but was exempt from the cataract assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Palifermin
Number analyzed (Participants) | 22 | 79
units on a scale
  Summary of difference from baseline in P | 0.01 (0.08) | 0.12 (0.40)
  Summary of difference from baseline in C | 0.14 (0.29) | 0.15 (0.28)
  Summary of difference from baseline in NO | 0.12 (0.26) | 0.35 (0.59)
Statistical Analysis 1: Comparison: Placebo vs Palifermin; Test type: Superiority or Other; Mean Difference (Net) = 0.023, 95% CI 2-sided [-0.134 to 0.181]

8. Secondary Outcome: Change From Baseline in Posterior Subcapsular (P), Cortical (C) Cataract and Nuclear Opalescence (NO) on the Lens Opacities Classification System III (LOCS III) Scale at Months 12.
Description: To study the change in cataract from baseline visit to months 12, regarding the three cataract main types: nuclear, cortical and posterior subcapsular measured on the Lens Opacities Classification System III (LOCS III) Scale. To assess the effect of palifermin on the incidence of cataract development or progression at Month 6 and Month 12 based on an increase of ≥ 0.3 in the Lens Opacities Classification System (LOCS III) score for Posterior Subcapsular cataract (P), Cortical Cataract (C) and Nuclear Opalescence (NO).
  The LOCS III is a standard system used for grading and comparison of cataract severity and type. The ophthalmologist uses a slit lamp for examining the lens of the eye. The classification evaluates: P,C and NO. NO is graded on a decimal scale of 0.1 to 6.9, based on a set of 6 standardized photographs. C and P are graded on a decimal scale of 0.1 to 5.9, based on a set of 5 standardized photographs each.
Time Frame: Months 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Palifermin
Number analyzed (Participants) | 22 | 79
units on a scale
  Summary of difference from baseline in P | 0.05 (0.12) | 0.25 (0.56)
  Summary of difference from baseline in C | 0.14 (0.25) | 0.22 (0.36)
  Summary of difference from baseline in NO | 0.12 (0.26) | 0.35 (0.59)
Statistical Analysis 1: Comparison: Placebo vs Palifermin; Test type: Superiority or Other; Mean Difference (Final Values) = 0.061, 95% CI 2-sided [-0.138 to 0.260]

9. Secondary Outcome: Incidence of a Decreased From Baseline in Best Corrected Visual Acuity (BCVA) as Measured by a Change of 10 Letters on the ETDRS (Early Termination Diabetic Retinopathy Study) at 4 Meters at Months 6
Description: To study if the treatment has effected on the visual acuity from baseline to months 6, by using Best Corrected Visual Acuity (BCVA) as measured by a Change of 10 Letters on the ETDRS (Early Termination Diabetic Retinopathy Study) at 4 Meters. To assess the effect of palifermin on the incidence of cataract development or progression at Month 6 and Month 12 based on an increase of ≥ 0.3 in the Lens Opacities Classification System (LOCS III) score for Posterior Subcapsular cataract (P), Cortical Cataract (C) and Nuclear Opalescence (NO).
Time Frame: Months 6
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | Placebo | Palifermin
Number analyzed (Participants) | 22 | 79
participants
  Incidence of decrease in letters read - Yes | 2 | 4
  Incidence of decrease in letters read - No | 15 | 48
  Subjects who discontinued at Month 6 | 5 | 27
Statistical Analysis 1: Comparison: Placebo vs Palifermin; Test type: Superiority or Other; Risk Difference (RD) = -3.689, 95% CI 2-sided [-21.641 to 14.264]

10. Secondary Outcome: Incidence of a Decreased From Baseline in Best Corrected Visual Acuity (BCVA) as Measured by a Change of 10 Letters on the ETDRS (Early Termination Diabetic Retinopathy Study) at 4 Meters at Months 12.
Description: To study if the treatment has effected on the visual acuity from baseline to months 12, by using Best Corrected Visual Acuity (BCVA) as measured by a Change of 10 Letters on the ETDRS (Early Termination Diabetic Retinopathy Study) at 4 Meters. To assess the effect of palifermin on the incidence of cataract development or progression at Month 6 and Month 12 based on an increase of ≥ 0.3 in the Lens Opacities Classification System (LOCS III) score for Posterior Subcapsular cataract (P), Cortical Cataract (C) and Nuclear Opalescence (NO).
Time Frame: Month 12
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | Placebo | Palifermin
Number analyzed (Participants) | 22 | 79
participants
  Incidence of decrease in letters read - Yes | 0 | 3
  Incidence of decrease in letters read - No | 14 | 49
  Subjects who discontinued at month 12 | 8 | 27
Statistical Analysis 1: Comparison: Placebo vs Palifermin; Test type: Superiority or Other; Risk Difference (RD) = 5.951, 95% CI 2-sided [-0.679 to 12.580]

11. Secondary Outcome: Incidence of Adverse Events and Laboratory Abnormalities
Description: Incidence of Adverse Events CTCAE grade 3 or higher reported
Time Frame: at Day 32
Measure: Number; unit: Participants
Arm/Group | Palifermin Before Only | Placebo | Palifermin Before and After
Number analyzed (Participants) | 111 | 57 | 109
Participants | 56 | 26 | 65

12. Secondary Outcome: Overall Survival
Description: Overall survival (OS) is based on death from any cause, not just the condition being treated, thus it picks up death from side effects of the treatment, and effects on survival after relapse.
Time Frame: During long-term follow up phase (maximum of 10 years)
Population: A total of 277 subjects were included in the Safety subset of the original study report (220 Palifermin and 57 placebo). Follow-up time for all subjects, defined as the date of randomization to the last known alive date. For subjects who were alive at the last contact the number of subjects for the palifermin group was 162 and for the placebo 47
Measure: Median (Inter-Quartile Range); unit: Months
Groups:
- Palifermin (Palifermin Before Only and, Before and After): Subjects to receive palifermin before-high dose chemotherapy (total 3 doses) and matched placebo after-high dose chemotherapy (total 3 doses) AND Subjects to receive palifermin before- and after-high dose chemotherapy (total of 6 doses)
Arm/Group | Palifermin (Palifermin Before Only and, Before and After) | Placebo
Number analyzed (Participants) | 220 | 57
Months | 50.6 [35.9 to NA] — Quartile 3 value is not available because a small number of participants died. | NA [44.1 to NA] — Median and quartile 3 values are not available because a small number of participants died.
Statistical Analysis 1: Comparison: Palifermin (Palifermin Before Only and, Before and After) vs Placebo; All comparisons for the long-term safety endpoints were based on the combined palifermin group (pre- and post- high dose chemotherapy and pre-high dose chemotherapy only) versus placebo (placebo over palifermin). Overall survival was analyzed using the Kaplan-Meier method. Kaplan-Meier estimates were provided together with the 95% confidence interval; Test type: Superiority or Other; p = 0.192, Log Rank; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.33 to 1.26]

13. Primary Outcome: Incidence of Cataract Development or Progression at Month 12.
Description: as for outcome 5
Time Frame: 12 months
Population: Of the 281 subjects who participated in the acute phase of the study a total of 101 subjects study were eligible for participation in the cataract assessment procedures, 22 in the placebo group and 79 in the palifermin group.
Measure: Number; unit: Participants
Arm/Group | Placebo | Palifermin
Number analyzed (Participants) | 22 | 79
Participants
  Yes | 4 [NA to NA] | 25 [NA to NA]
  No | 10 [NA to NA] | 27 [NA to NA]
  Missing | 8 [NA to NA] | 27 [NA to NA]
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 17.417, 95% CI 2-sided [-11.086 to 45.919]

14. Secondary Outcome: Progression Free Survival
Description: Progression-free survival (PFS) is the length of time during and after the treatment during which the disease being treated does not get worse. In this study the event for Progression-free survival was death from all causes or disease progression. Time to each event was defined as the time elapsed between the date of the first dose of investigational product, and the date of the given event.
Time Frame: During long-term follow up phase (maximum of 10 years)
Population: as for outcome 12
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Palifermin (Palifermin Before Only and, Before and After) | Placebo
Number analyzed (Participants) | 220 | 57
Months | 15.1 [8.4 to 24.0] | 18.3 [11.9 to 27.5]
Statistical Analysis 1: Comparison: Palifermin (Palifermin Before Only and, Before and After) vs Placebo; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.236, Log Rank; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.55 to 1.16]

15. Secondary Outcome: Time Death or Disease Progression
Description: For the analysis of time to disease progression, competing risks time-to-event analysis was used, since a subject destined to develop disease progression could die from unrelated causes before the disease progression event takes place. Kaplan-Meier survival estimates, with death due to other causes than progression considered as a competing risk, were provided: event rate at 3 month intervals, with 95% confidence interval, the number of subjects at risk at the beginning of the time period, and the number of events of interest.
Time Frame: During long-term follow up phase (maximum of 10 years)
Population: as for outcome 12
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Palifermin (Palifermin Before Only and, Before and After) | Placebo
Number analyzed (Participants) | 220 | 57
months | 15.1 [8.4 to 24.0] | 18.3 [11.9 to 27.5]
Statistical Analysis 1: Comparison: Palifermin (Palifermin Before Only and, Before and After) vs Placebo; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.372, Log Rank; Hazard Ratio, log = 0.84, 95% CI 2-sided [0.58 to 1.23]

16. Secondary Outcome: Incidence of Second Primary Malignancies or Other Malignancies
Description: All comparisons for the long-term safety endpoints were based on the combined palifermin group versus placebo (placebo over palifermin). Incidence of new or secondary malignancies by treatment group was provided (incidence of new or secondary malignancies at the follow-up visit - yes, no, no assessment -, and number of subjects with new or secondary malignancies, per type of malignancies). The long-term safety evaluations were summarized for the subgroups defined by the factors used for randomization using descriptive statistics.
Time Frame: During long-term follow up phase (maximum of 10 years)
Population: total of 277 subjects were included in the Safety subset of the original study report (220 Palifermin and 57 placebo). Follow-up time for all subjects, defined as the date of randomization to the last known alive date. For subjects who were alive at the last contact the number of subjects for the palifermin group was 162 and for the placebo 47.
Measure: Number; unit: participants
Arm/Group | Palifermin (Palifermin Before Only and, Before and After) | Placebo
Number analyzed (Participants) | 220 | 57
participants | 1 | 6

ADVERSE EVENTS:
Time Frame: Adverse Events were collected for a period of up to 222 days.
Groups:
- Palifermin Before Only: Subjects to receive palifermin before-high dose chemotherapy (total 3 doses) and matched placebo after-high dose chemotherapy (total 3 doses). A total of 109 subjects were randomized to treatment and 107 received at least one dose of study treatment. Due to protocol deviations 4 patients randomized to Palifermin Before and After group were included Palifermin Before Only group and therefore a total of 111 subjects were included in this safety analysis set.
- Palifermin Before and After: Subjects to receive palifermin before- and after-high dose chemotherapy (total of 6 doses). A total of 115 subjects were randomized to treatment and 113 received at least one dose of study treatment. Due to protocol deviations additional 4 patients randomized to Palifermin Before and After group were included Palifermin Before Only group and therefore a total of 109 subjects were included in this safety analysis set.
Arm/Group | Palifermin Before Only | Placebo | Palifermin Before and After
Serious Adverse Events (participants affected / at risk) | 13/111 | 3/57 | 18/109
Other Adverse Events (participants affected / at risk) | 110/111 | 56/57 | 109/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Palifermin Before Only (N=111) | Placebo (N=57) | Palifermin Before and After (N=109)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 1 | 1
Catheter related infection (Infections and infestations) | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Edema (General disorders) | 0 | 0 | 1
Epiglottitis (Infections and infestations) | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 1
Face oedema (General disorders) | 0 | 0 | 1
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 1
Graft complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1
Infection (Infections and infestations) | 1 | 0 | 1
Intervertebral discitis (Infections and infestations) | 1 | 0 | 0
Mediastinitis (Infections and infestations) | 0 | 0 | 1
Melanodermia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 2
Pneumonia primary atypical (Infections and infestations) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 1 | 1
Septic shock (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Tongue discolouration (Gastrointestinal disorders) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0
Weight decreased (Investigations) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Palifermin Before Only (N=111) | Placebo (N=57) | Palifermin Before and After (N=109)
Abdominal pain (Gastrointestinal disorders) | 12 | 8 | 9
Abdominal pain upper (Gastrointestinal disorders) | 13 | 8 | 11
Anemia (Blood and lymphatic system disorders) | 19 | 7 | 17
Anorexia (Metabolism and nutrition disorders) | 10 | 7 | 12
Anxiety (Psychiatric disorders) | 6 | 3 | 7
Asthenia (General disorders) | 8 | 6 | 14
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 5 | 6
Constipation (Gastrointestinal disorders) | 23 | 11 | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 3 | 7
Diarrhoea (Gastrointestinal disorders) | 80 | 42 | 81
Dysgeusia (Nervous system disorders) | 7 | 3 | 6
Dyspepsia (Gastrointestinal disorders) | 9 | 1 | 9
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 5
Edema (General disorders) | 13 | 9 | 16
Edema peripheral (General disorders) | 13 | 4 | 17
Erythema (Skin and subcutaneous tissue disorders) | 20 | 4 | 26
Fatigue (General disorders) | 13 | 9 | 11
Febrile neutropenia (Blood and lymphatic system disorders) | 16 | 12 | 19
Hypertension (Vascular disorders) | 15 | 2 | 11
Hypokalemia (Metabolism and nutrition disorders) | 20 | 7 | 16
Hypotension (Vascular disorders) | 7 | 3 | 7
Infection (Infections and infestations) | 6 | 2 | 7
Insomnia (Psychiatric disorders) | 10 | 7 | 11
Leukopenia (Blood and lymphatic system disorders) | 16 | 4 | 12
Nausea (Gastrointestinal disorders) | 87 | 44 | 77
Neutropenia (Blood and lymphatic system disorders) | 18 | 5 | 13
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 15 | 9 | 15
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 6 | 15
Pyrexia (General disorders) | 48 | 22 | 47
Rash (Skin and subcutaneous tissue disorders) | 24 | 12 | 41
Tachycardia (Cardiac disorders) | 2 | 2 | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 22 | 9 | 19
Vomiting (Gastrointestinal disorders) | 46 | 25 | 44
Weight increased (Investigations) | 4 | 7 | 5
Headache (Nervous system disorders) | 18 | 6 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits sponsor a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Sponsor may remove confidential information, but authors have final control and approval of publication content. For multi-center studies, investigator agrees not to publish any results before the first multi-center publication.